CLINICAL TRIAL: NCT04047433
Title: The Occurrence of Single Nucleotide Polymorphism Among Women Who Experienced Obstetric Anal Sphincter Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Eyal Rom, MD, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 0091-18-EMC
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Delivery, Obstetric
MeSH Terms: interventions — Mass Screening; Polymorphism, Single Nucleotide; Exome Sequencing

STUDY DESIGN:
Intervention Model Description: two arms -
  1. with external anal sphincter injury
  2. without injury both will go through genetic screening test the arm with the external anal sphincter injury will also be tested for advanced genetic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- women with external anal sphincter injury (Experimental): The study cohort will be composed of women undergoing vaginal delivery and diagnosed with external anal sphincter injury after a vaginal delivery.
  Interventions: Genetic: screening for single nucleotide polymorphism; Genetic: whole exome sequencing
- women without external anal sphincter injury (Experimental): The control group will be women who had a vaginal delivery without any clinically apparent perineal laceration
  Interventions: Genetic: screening for single nucleotide polymorphism

INTERVENTIONS:
Genetic: screening for single nucleotide polymorphism — samples from both arms will be tested for a set of single nucleotide polymorphism
Genetic: whole exome sequencing — samples from arm #1 (women with external anal sphincter) will be tested for identifying specific genetic mutation
  Arms: women with external anal sphincter injury

SUMMARY:
Single-nucleotide polymorphisms (SNP's) in connective tissue components are associated with increased risk of pelvic organ prolapse (POP). The investigators expect to find a difference in SNP's frequency between women who had Obstetric anal sphincter injuries (OASIS) and in the healthy population. The fact that pelvic organ prolapse (POP) and OASIS occurs in the same anatomic region and the well-known association between few SNP's and the risk for POP, suggests for a common pathophysiology.

DETAILED DESCRIPTION:
The perineum consists of skin, muscles and connective tissue. A connective tissue disorder related to POP has been reported in biochemical and molecular studies. OASIS are considered a severe complication of vaginal delivery that may lead to a great deal of morbidity. Familial history is known as a risk factor for OASIS. Currently, there is no established genetic link between connective tissue components and OASIS. Therefore, the investigators assume that studying the genetic predisposition factors of women who experience OASIS, might generate a stronger tool to predict severe occurrence of vaginal laceration. It may also help to consult women before vaginal delivery about the risk of OASIS.

The aim of this study is to find an association between genetic variation and increased risk for OASIS.

ELIGIBILITY:
Inclusion Criteria:

* Women with severe external anal sphincter injury during first vaginal delivery
* Healthy women undergoing vaginal delivery without any clinically apparent perineal laceration

Exclusion Criteria:

* Women with known metabolic or connective-tissue disorder (e.g., Ehlers-Danlos syndrome).
* Women with known neurologic disorder
* Women undergoing episiotomy cut or assisted delivery (e.g., vacuum or forceps delivery)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
difference in the frequency of of Single-nucleotide polymorphisms | through study completion, an average of 2 years
  difference in the relative frequency of Single-nucleotide polymorphisms between women with external anal sphincter injury that occurs during vaginal delivery and those without it.

SECONDARY OUTCOMES:
genetic mutation | through study completion, an average of 2 years
  specific genetic mutation among women with external anal sphincter injury that occurs during vaginal delivery

CONTACTS AND LOCATIONS:
Overall Officials: Hedi Raischer, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel, Israel

IPD SHARING:
Plan to Share IPD: No